CLINICAL TRIAL: NCT07187297
Title: A Prospective Controlled Study to Evaluate the Safety and Effectiveness of Thermage® FLX Radiofrequency Treatment to Improve Lines and Wrinkles and to Lift and Tighten Lax Tissue in the Neck, Abdomen, Upper Arms, and Face
Brief Title: A Prospective Controlled Study to Evaluate the Safety and Effectiveness of Thermage® FLX Radiofrequency Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: TM-PAS-NAPAC-2025-001
Record Dates: First submitted 2025-09-18; First posted 2025-09-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Wrinkle; Lax Skin; Lines Skin
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Arm (Active Comparator): Treated with Thermage FLX device at day 90
  Interventions: Device: Thermage FLX
- Treatment Arm (Experimental): Treated with Thermage FLX device at day 1
  Interventions: Device: Thermage FLX

INTERVENTIONS:
Device: Thermage FLX — The Thermage FLX System ('System') is a monopolar, capacitively coupled radiofrequency System designed for use in non-invasive dermatological procedures

SUMMARY:
A prospective, 180-day, randomized, multicenter, independent blinded evaluators, controlled study of treatment with the Thermage FLX System

DETAILED DESCRIPTION:
Study to be conducted at approximately 10 study centers, enrolling a total of 164 participants in North America (US and Canada) and China. Approximately 6 months (26 weeks) Purpose is to demonstrate superiority of treatment with the Thermage FLX System compared to untreated control for the improvement of:

Lines and wrinkles of the neck and face Skin laxity of the neck, abdomen, upper arms, and face and evaluate safety and tolerability of treatment with the Thermage FLX System compared to the untreated control arm.

ELIGIBILITY:
Inclusion Criteria:

* Be an adult female or male, ≥30 - ≤60 years of age.

Have mild-to-moderate skin laxity of the neck, abdomen, upper arms, and/or face, and/or mild-to-moderate lines and/or wrinkles of the neck and/or face assessed as follows:

Neck:

Mild-to-moderate neck skin laxity as defined by a score of 1 to 6 on the 10-point Facial Laxity Rating Scale (scored 0-9)

Mild-to-moderate neck wrinkles as defined by a score of 1 to 6 on the 10-point Fitzpatrick Wrinkle Scale (scored 0-9)

Abdomen:

Mild-to-moderate abdomen skin laxity as defined by a score of 1 or 2 on a 4-point Abdominal Laxity Scale (scored 0-3)

Upper arms:

Mild to moderate upper arms skin laxity as defined by grade 2 or 3 on the 5-grade IBSA Inner Upper Arm Laxity Scale

Face:

Mild-to-moderate facial skin laxity as defined by a score of 1 to 6 on the 10-point Facial Laxity Rating Scale (scored 0-9)

Mild-to-moderate facial wrinkles as defined by a score of 1 to 6 on the 10-point Fitzpatrick Wrinkle Scale (scored 0-9)

Females of childbearing potential must have a negative urine pregnancy test. Females who have experienced menarche and who are not postmenopausal (either confirmed via FSH testing or who have not menstruated for 2 years or more without an alternative medical cause) or surgically sterile will be considered of childbearing potential.

Females of childbearing potential must agree to use an acceptable method of birth control for the duration of the study. Acceptable methods of birth control are oral and other systemic contraceptives, condoms only, intrauterine device, double-barrier methods, bilateral tubal ligation, partner vasectomy, and abstinence.

Have no clinically abnormal findings based on the medical history as determined by the study investigator.

Be able to follow the study instructions, be available on the specific required study visit days, and be willing to complete all study visit procedures and assessments.

Understand the research nature of this study and sign an informed consent document prior to the performance of any study-specific procedure or assessment.

Agree to not undergo excluded procedures (i.e., energy-based device treatments, injectables, or plastic surgery) on the study treatment areas for the duration of study.

Participant has a body mass index (BMI) ≤30.

Exclusion Criteria:

* Participant is pregnant or breast feeding or trying to become pregnant for 3 months prior to the screening visit or during the study.

Participant has given birth within 3 months prior to the screening visit.

Participant has an anticipated need for procedures, surgery, overnight hospitalization, or other events that would prevent the participant from making the required visits during the study.

Participant has a pacemaker, internal defibrillator, or other implanted electronic device.

Participant has an implant in the target treatment zone(s).

Participant has had radiation therapy in the target treatment zone(s).

Participant has had 1 or more prior cosmetic procedures in the target treatment zone(s) including:

Thermage or any energy-based device procedure, derm abrasion, or chemical peel on any treatment area within 6 months prior to the screening visit.

Short-acting neurotoxins within 6 months prior to the screening visit.

Long-acting neurotoxins within 9 months prior to the screening visit.

Hyaluronic acid filler ≤1 year prior to the screening visit.

Semi-permanent or permanent fillers at any time prior to the screening visit.

Plastic surgery within 1 year prior to the screening visit.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 90 days
  Proportion of participants with any improvement on iGAIS at Day 90 as assessed by independent blinded evaluators.

SECONDARY OUTCOMES:
Secondary Endpoint | 180 days
  Proportion of participants with any improvement on iGAIS, Fitzpatrick Wrinkle Scale, Facial Laxity Rating Scale, IBSA Inner Upper Arm Laxity Scale, Abdominal Laxity Scale at Day 90 and 180.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Square Laser Dermatology, New York, New York, United States